CLINICAL TRIAL: NCT04780399
Title: Efficacy and Safety of Yangxue Qingnao Pills in the Treatment of Mild to Moderate Alzheimer's Disease:a Multicenter, Randomized, Double-blind, Placebo-controlled, Phase II Clicnial Trial
Brief Title: Efficacy and Safety of Yangxue Qingnao Pills in the Treatment of Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, Vice president, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2020-03-BDY-12-V02
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease; Yangxue Qingnao Pills; Randomized
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yangxue Qingnao pills high dose group (Experimental): Yangxue Qingnao pills 7.5 g per time,2 times per day.
  Interventions: Drug: Yangxue Qingnao pills
- Yangxue Qingnao pills lower dose group (Experimental): Yangxue Qingnao pills 5 g per time,2 times per day, and placebo identified to Yangxue Qingnao pills 2.5 g per time, 2 times per day.
  Interventions: Drug: Yangxue Qingnao pills
- Placebo group (Placebo Comparator): Placebo identified to Yangxue Qingnao pills 7.5 g per time,2 times per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yangxue Qingnao pills — 72 subjects in the Yangxue Qingnao pills group take 7.5g of Yangxue Qingnao pills each time, twice a day, 0.5 hours after breakfast and dinner, taking with warm water.
  Arms: Yangxue Qingnao pills high dose group
Drug: Yangxue Qingnao pills — 72 subjects in the Yangxue Qingnao pills group take 5g of Yangxue Qingnao pills and 2.5g placebo identified to Yangxue Qingnao pills each time, twice a day, 0.5 hours after breakfast and dinner, taking with warm water.
  Arms: Yangxue Qingnao pills lower dose group
Drug: Placebo — 72 subjects in the placebo group take 7.5g placebo identified to Yangxue Qingnao pills each time, twice a day, 0.5 hours after breakfast and dinner, taking with warm water.
  Arms: Placebo group

SUMMARY:
As a traditional Chinese medicine compound, Yangxue Qingnao Pills is proven to have beneficial effects on learning and memory ability in animal models of Alzheimer's disease(AD). The purpose of the study is to evaluate the efficacy and safety of Yangxue Qingnao Pills on patients with mild to moderate AD. This phase II randomized, double-blind, parallel controlled trial include a 2 weeks run-in period, and a 48 weeks double-blind treatment period of after randomization. Participants will be randomly allocated to Yangxue Qingnao pills high dose group (7.5 g per time,2 times per day) ; and Yangxue Qingnao pills low dose group (5 g per time,2 times per day), or placebo group. The outcome measures include general cognitive function, ability of daily living, and behavioural and psychological symptoms in AD patients.

DETAILED DESCRIPTION:
Yangxue Qingnao pills is a traditional Chinese herbal medicine, which is composed of Angelicae Sinensis Radix , Chuanxiong Rhizoma , Paeoniae Radix Alba, Rehmannia glutinosa, Uncaria macrophylla Wall, Caulis spatholobi, Spica Prunellae, Catsia tora Linn , Mater Margarita, Corydalis ambigua and Asarum sieboldii. The function of Yangxue Qingnao pills is nourishing blood and calming liver, promoting blood circulation and dredging collaterals in Chinese traditional medicine theory. This study is a 48-weeks, multicenter, randomized, double-blind, parallel controlled phase II trial being carried out in China. The study population includes mild to moderate Alzheimer's disease (planned a total of 216) aged 65-85 in both gender. Participants will be randomly allocated to Yangxue Qingnao pills high dose group (7.5 g per time,2 times per day) ; and Yangxue Qingnao pills low dose group (5 g per time,2 times per day), or placebo group for a 48-weeks double-blind treatment period. The primary outcome measure is change from baseline in the Alzheimer's Disease Assessment Scale- Cognition Subscale (ADAS-cog) and the clinical dementia rating scale. The secondary outcomes are changes from baseline in the Mini-Mental State Examination(MMSE), Alzheimer's Disease Cooperative Study-Activities of Daily Living scale (ADCS-ADL/24) and Neuropsychiatric Inventory. Besides, the blood biomarkers including Aβ42, Aβ40, T-tau, P-tau181, NfL, TOM1, IL-1R1,IL-1b, IL-6, IL-8, TNF-a, FB, FH, sCR1, MCP-1, eotaxin-1, Ach, ChEI and the hippocampal volume on MRI. Safety is being assessed by observing side effects and adverse reaction during the entire treatment period. Statistical analysis will be conducted according to per-protocol population and intend-to-treat population and the safety will be analyzed in safety set.

ELIGIBILITY:
Inclusion Criteria:

Patients, Chinese speaking, in both gender are eligible to be included in the study only if they meet all of the following criteria:

1. Meets NIA/AA core clinical criteria for probable AD;
2. The body weight is between 45-90kg;
3. Aged ≥ 65 and ≤ 85 years old;
4. Mild to moderate stage of AD, defined as( MMSE score of 15 through 26) at baseline;
5. Has had an MRI scan performed at baseline that has confirmed with a diagnosis of AD, Medial temporal atrophy scale (MTA) is used for routine assessment of the medial temporal lobe, and the MTA score need ≥1.5 (adjusted by age: 65-74 years ≥ 1.5 points, 75-84 years old ≥ 2.0 points);
6. Has a PIB-PET scan or CSF result consistent with the presence of amyloid pathology at screening;
7. And the patients must have adequate vision and hearing to participate in study assessments; has normal swallowing function, and can complete the medication;
8. Have a stable caregiver;
9. Can read simple articles and write simple sentences;
10. Informed consent, signed informed consent by legal guardian.

Exclusion Criteria:

Patients who confirmed with any of the following excluding criteria conditions were not enrolled for the study:

1. Early-onset Alzheimer disease (oneset at <65 years of age) and moderate to severe AD dementia (MMSE 14-0);
2. Evidence of other reasons caused cognitive impairment, like vascular dementia, frontotemporal dementia, Parkinson's disease dementia, Lewy body dementia, Huntington's disease, subdural hematoma, communicating hydrocephalus, brain tumor, thyroid disease, vitamin deficiency Or other diseases that may cause cognitive impairment, or serious brain infections (including neurosyphilis, meningitis or encephalitis), etc.;
3. There are unstable mental disorders, including major depression (HAMD≥17), severe anxiety disorder (HAMA≥12 points), bipolar disorder, schizophrenia, etc.;
4. History of drug or alcohol abuse in the past 5 years;
5. Other uncontrolled chronic illnesses, such as severe arrhythmia (ventricular rate <60 beats/min or >100 beats/min, or patients with myocardial infarction within 3 months before participating in the trial, or severe heart failure (NY classification III and IV), or severe abnormal blood pressure, systolic blood pressure ≤90mmHg or ≥180mmHg;
6. Severe liver or kidney dysfunction (alanine aminotransferase or aspartate transaminase was more than 1.5 times the upper limit of normal, or serum creatinine was more than the upper limit of normal);
7. A history of taking cholinesterase inhibitors, memantine, or proprietary Chinese medicines with clear nootropic effects within the past 1 month;
8. Has received medications that affect the central nervous system (CNS), except treatments for AD for less than 4 weeks; that is, doses of chronic medications that affect the CNS should be stable for at least 4 weeks;
9. One of the following manifestations on cranial MRI:> 4 cerebral microhemorrhages, evidence of a prior macrohemorrhage, > 3 lacunar infarcts over 10 mm each, any cortical infarct over 10 mm, or any other clinically significant finding (e.g., any lesion that may account for their cognitive impairment, including but not limited to brain tumor, severe white matter disease with a rating of 3 on the Fazekas scale for WM lesions ,arteriovenous malformation, cavernous hemangioma, or any infarct in a strategic subcortical location);
10. History of hypersensitivity to the treatment drugs;
11. Participate in other clinical study within the last 30 days;
12. Has metal (ferromagnetic) implants, or a cardiac pacemaker and other conditions that could not undergo MRI scan;
13. or other conditions that, in the investigator's opinion, could interfere with the analyses of safety and efficacy in this study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale- Cognition Subscale (ADAS-cog) | Change from baseline ADAS-cog score at Week 48
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale test is one of the most frequently used tests to measure cognition in research studies and clinical trials for new drugs and other interventions.The ADAS-Cog consists of 11 parts and takes approximately 30 minutes to administer.The test administrator adds up points for the errors in each task of the ADAS-Cog for a total score ranging from 0 to 70. The greater the dysfunction, the greater the score. A score of 70 represents the most severe impairment and 0 represents the least impairment.
Clinical dementia rating scale-sum box(CDR-SB) | Change from baseline CDR-SB score at Week 48
  The Clinical Dementia Rating Scale (CDR) is a global assessment instrument that yields global and Sum of Boxes (CDR-SB) scores, with the global score regularly used in clinical and research settings to stage dementia severity. The CDR-SB score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18. Higher score means severe global cognition impairment.

SECONDARY OUTCOMES:
Mini-Mental State Examination(MMSE) | Change from baseline MMSE score at Week 48
  TThe Mini-Mental Status Examination offers a quick and simple way to quantify cognitive function and screen for cognitive loss. It tests the individual's orientation, attention, calculation, recall, language and motor skills. It takes ~ 5-10 minutes to administer The range for the total MMSE score is 0 to 30, higher score means better cognition.
Neuropsychiatric Inventory(NPI) | Change from baseline NPI score at Week 48
  The NPI is a semistructured clinician interview of caretakers in which the severity and frequency of disturbance in 12 symptom domains is rated
Alzheimer's Disease Cooperative Study-Activities of Daily Living scale (ADCS-ADL/23) | Change from baseline ADCS-ADL/23 score at Week 48
  The Alzheimer's Disease Cooperative Study (ADCS) tested 23-item version (ADCS-ADL/23) includes more complex ADL for the assessment of mild to moderate AD, such as reading books or magazines, pastime activities, or household chores. Ratings take about 20 minutes and are based on information obtained from the patient and caregiver. The scores range from 0 to 78, higher scores indicating less functional impairment.

OTHER OUTCOMES:
Blood biomarkers including Aβ42, Aβ40, T-tau, P-tau181, NfL, TOM1, IL-1R1,IL-1b, IL-6, IL-8, TNF-a, FB, FH, sCR1, MCP-1, eotaxin-1, Ach, ChEI | Change from baseline of Aβ42, Aβ40, T-tau, P-tau181, NfL, TOM1, IL-1R1,IL-1b, IL-6, IL-8, TNF-a, FB, FH, sCR1, MCP-1, eotaxin-1, Ach, ChEI at Week 48
Hippocampus volume with MRI | Change of hippocampus volume with MRI after 48 weeks'treatment from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, MD,PhD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital ,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China